CLINICAL TRIAL: NCT04280809
Title: Postoperative Analgesic and Anti-inflammation Effects of Low-level Laser Therapy After Surgical Removal of Impacted Lower Third Molar
Brief Title: Effects of Low-level Laser Therapy After Surgical Removal of Impacted Lower Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Le Thanh Thai Ha, Faculty of Odonto-Stomatology, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NT62 72 28 01
Record Dates: First submitted 2020-02-14; First posted 2020-02-21 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Facial Swelling; Pain; Trismus
MeSH Terms: conditions — Pain; Trismus | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser (Experimental): Subsequently to the suture, laser was applied in the right or left side randomly on each patient, according to a sheet of randomization. GaAlAs laser (AMD Picasso, Dentsply Sirona, York, Pennsylvania, USA) with a wavelength of 810 nm was placed intraorally, at a distance of 1 cm in the position of the extracted tooth socket and circling in a 2 cm - diameter area. The power applied was 0.5 ± 20% W, continuously for 30 s. The total real energy released was 12.8 J and the real energy density applied was 4 J/cm2.
  Interventions: Device: GaAlAs laser
- Non-laser (No Intervention): Every patient, on the control side, the same handpiece was applied intraorally, but laser was not activated

INTERVENTIONS:
Device: GaAlAs laser — GaAlAs laser (AMD Picasso, Dentsply Sirona, York, Pennsylvania, USA) with a wavelength of 810 nm was placed intraorally, at a distance of 1 cm in the position of the extracted tooth socket and circling in a 2 cm - diameter area. The power applied was 0.5 ± 20% W, continuously for 30 s. The total real energy released was 12.8 J and the real energy density applied was 4 J/cm2. Each patient was irradiated 3 times consecutively right after surgery, day 1 and day 2 after surgery
  Arms: Laser

SUMMARY:
Goal: The aim of this study was to evaluate the effects of low-level laser (LLL) after surgical removal of impacted lower third molars (ILTM).

DETAILED DESCRIPTION:
Goal: The aim of this study was to evaluate the effects of low-level laser (LLL) after surgical removal of impacted lower third molars (ILTM), including pain level, postoperative facial swelling, trismus and non-stimulated saliva secretory immunoglobulin A (sIgA).

ELIGIBILITY:
Inclusion Criteria:

* had two impacted lower third molars symmetrically in the same position as the classifications of Pell- Gregory and Winter diagnosed by 2D panoramic radiography

Exclusion Criteria:

* Patients with systemic diseases such as cardiovascular disease, hypertension, diabetes mellitus, pregnant, local infections
* refused to participate in the study
* patients who did not follow-up visit would be excluded

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Pain degree | at 2 hours after stopping the feeling of numbness lips
  Likert scale
Pain degree | at 4 hours after stopping the feeling of numbness lips
  Likert scale
Pain degree | at 6 hours after stopping the feeling of numbness lips
  Likert scale
Pain degree | at 24 hours after surgery
  Likert scale
Pain degree | at 48 hours after surgery
  Likert scale
Face swelling degree | on first day after surgery
  Mark indelibly on the skin of points used to record the preoperative swelling level based on benchmarks A, B, C, D. A was the external canthus of the eye, B was the Gonion, C was the lip-commissure and D was the lowest point of the earlobe. The degree of face swelling was determined by using measuring tape (rounded to the nearest millimeter line): vertically from the external canthus of the eye to the Gonion (segment AB) and horizontally: from earlobe to the lip-commissure (CD segment). To evaluate generally face swelling, we computed the swelling area (mm2) approximately by the formula AB*CD/2
Face swelling degree | on second day after surgery
  Mark indelibly on the skin of points used to record the preoperative swelling level based on benchmarks A, B, C, D. A was the external canthus of the eye, B was the Gonion, C was the lip-commissure and D was the lowest point of the earlobe. The degree of face swelling was determined by using measuring tape (rounded to the nearest millimeter line): vertically from the external canthus of the eye to the Gonion (segment AB) and horizontally: from earlobe to the lip-commissure (CD segment). To evaluate generally face swelling, we computed the swelling area (mm2) approximately by the formula AB*CD/2
Trismus degree | on day 1 postoperatively
  measuring the distance between the mesial angle of the central incisors of the upper and lower (maximum oral aperture, MOA) of the patient with a caliper
Trismus degree | on day 2 postoperatively
  measuring the distance between the mesial angle of the central incisors of the upper and lower (maximum oral aperture, MOA) of the patient with a caliper
sIgA concentration | the second day after surgery
  Firstly, the saliva sample was centrifuged for 10 minutes, speed 3000 rpm, at 40 degrees Celsius. After eliminating oral mucosa cells, red blood cells, the 500 µl of the sample solution was added 5 µl proteolytic inhibitor to avoid cleavage of the sIgA antibodies in the sample to be investigated. The sample was vibrated with a vortex vibrator for 20 seconds and stored in -80°C. After collecting enough samples, the samples were performed the Elisa sandwich procedure according to the standard instructions of Kit Elisa Elabscience Human Secretory IgA (Elabscience Biotechnology, Houston, Texas, US) using Elisa IRE 96 SFRI Kit reader 450nm (SFRI, Saint-Jean-d'Illac, France)

OTHER OUTCOMES:
Face swelling degree | before surgery
  Mark indelibly on the skin of points used to record the preoperative swelling level based on benchmarks A, B, C, D. A was the external canthus of the eye, B was the Gonion, C was the lip-commissure and D was the lowest point of the earlobe. The degree of face swelling was determined by using measuring tape (rounded to the nearest millimeter line): vertically from the external canthus of the eye to the Gonion (segment AB) and horizontally: from earlobe to the lip-commissure (CD segment). To evaluate generally face swelling, we computed the swelling area (mm2) approximately by the formula AB*CD/2
sIgA concentration | before the surgery
  Firstly, the saliva sample was centrifuged for 10 minutes, speed 3000 rpm, at 40 degrees Celsius. After eliminating oral mucosa cells, red blood cells, the 500 µl of the sample solution was added 5 µl proteolytic inhibitor to avoid cleavage of the sIgA antibodies in the sample to be investigated. The sample was vibrated with a vortex vibrator for 20 seconds and stored in -80°C. After collecting enough samples, the samples were performed the Elisa sandwich procedure according to the standard instructions of Kit Elisa Elabscience Human Secretory IgA (Elabscience Biotechnology, Houston, Texas, US) using Elisa IRE 96 SFRI Kit reader 450nm (SFRI, Saint-Jean-d'Illac, France)

CONTACTS AND LOCATIONS:
Overall Officials: Ly TB Nguyen, PhD, Study Director — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Faculty of Odonto-Stomatology, Ho Chi Minh City, Dictrict 5, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le HT, Huynh NC, Nguyen-Ho QA, Nguyen TT, Le SH, Nguyen LT. Effect of Photobiomodulation Therapy on Reducing Acute Pain and Inflammation Following Surgical Removal of Impacted Mandibular Third Molars: A Randomized, Split-Mouth Clinical Trial. Photobiomodul Photomed Laser Surg. 2022 Apr;40(4):245-251. doi: 10.1089/photob.2021.0110. Epub 2022 Mar 29. PMID 35353636